CLINICAL TRIAL: NCT06923696
Title: Evaluating the Effects of Low FODMAP and Gluten-Free Diet on Nutritional Status, Quality of Life, and Gastrointestinal Symptoms in Irritable Bowel Syndrome (IBS)
Brief Title: Low FODMAP Diet and Gluten Free Diet in IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuh Naci Yazgan University (Other)
Responsible Party: Principal Investigator, Aslı Gizem Çapar, asst.prof., Nuh Naci Yazgan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: nuhnacıyazgan
Record Dates: First submitted 2024-03-26; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: IBS - Irritable Bowel Syndrome; Diet, Healthy; Elimination Disorder With Fecal Symptoms
Keywords: IBS; diet therapy; gluten-free diet; fodmap diet; life quality
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gluten free diet group (Experimental): Gluten-free diet therapy was implemented for 1 month
  Interventions: Behavioral: Diet therapy
- LOW FODMAP diet group (Experimental): Low FODMAP diet therapy was implemented for 1 month
  Interventions: Behavioral: Diet therapy

INTERVENTIONS:
Behavioral: Diet therapy — One of the groups will follow a gluten-free diet therapy, while the other will follow a LOW FODMAP diet.

SUMMARY:
The data of the research will be collected from patients who have applied to the Gastroenterology Polyclinic of Kayseri City Hospital or have previously been diagnosed with Irritable Bowel Syndrome (IBS). The data will be collected through face-to-face interviews using a questionnaire form. Participation in the study is entirely voluntary, and participants have the right to withdraw from the research at any time if they wish.

The general flowchart of the research is shown in Figure 1.

Figure 1. Flowchart of the Research

Patients with IBS applying to the Gastroenterology Polyclinic:

According to Rome IV criteria, individuals aged between 19-64, with BMI >18.5 and <29.9 kg/m2, non-cancerous, not using probiotics in the last month, and not following a gluten-free diet.

Interview Group 1: Low FODMAP diet Group 2: Gluten-free diet

Socio-demographic characteristics, general dietary habits, level of physical activity, anthropometric measurements, body composition analysis, IBS-SSS, IBS-QOL, IBS-VAS, Bristol Stool Scale, 24-hour retrospective food consumption record, Food Frequency Questionnaire.

Second Interview (after 4 weeks)

Anthropometric measurements, body composition analysis, IBS-SSS, IBS-QOL, IBS-VAS, Bristol Stool Scale, 3-day retrospective food consumption record.

DETAILED DESCRIPTION:
Survey Form The survey form administered to all participants in the study will include sociodemographic characteristics, information on general dietary habits (19 questions), physical activity (2 questions), and diagnostic information related to the disease (9 questions). Information on additional methods participants resort to alleviate their IBS symptoms (alternative treatments and dietary supplements such as fiber, prebiotics, probiotics, aloe vera, peppermint oil) will also be included in the survey.

Anthropometric Measurements Anthropometric measurements and body composition of the participants will be determined by the researcher after the diagnosis of IBS and before initiating any dietary intervention, as well as after a 4-week dietary intervention.

Body weight: The participants' body weight will be measured using the TANITA MC-780 model with minimal clothing and without shoes.

Height: Height measurement will be taken while the feet are together and the head is in the Frankfort plane (ear canal and bottom of the eye socket aligned horizontally, with the gaze parallel to the ground).

Body mass index (BMI): BMI will be calculated by dividing body weight in kilograms by the square of height in meters. BMI will be evaluated according to the classification provided by the World Health Organization (WHO). According to this classification, individuals with BMI <18.5 kg/m² are considered "underweight," those with BMI 18.5-24.9 kg/m² are considered "normal," individuals with BMI 25.0-29.9 kg/m² are classified as "overweight," those with BMI 30.0-34.9 kg/m² are considered "obese class 2," and those with BMI >40 kg/m² are considered "obese class 3." Waist circumference: Waist circumference will be measured using a non-stretchable tape measure at the midpoint between the lower rib and the iliac crest. Waist circumference will be evaluated according to the WHO classification, considering waist circumference greater than 102 cm in men and greater than 88 cm in women as high risk for metabolic complications.

Hip circumference: Hip circumference measurement will be taken while the participant stands on their left side, using a non-stretchable tape measure parallel to the ground at the highest point.

Dietary Intake Record To determine the energy and nutrient intake of individuals, detailed dietary intake records will be obtained retrospectively for 24 hours during the initial interview, and for 3 days during the second and final interviews. Standard recipes will be used to determine the portion sizes and quantities of consumed foods. The average daily energy and nutrient intake of individuals will be calculated using the Nutrition Information System computer software package. The adequacy of energy and nutrient intake relative to age and gender will be calculated based on the Turkish Dietary Guidelines , and the average percentage of meeting dietary requirements will be determined.

Food Frequency Consumption To assess changes in the dietary intake status of participants before and after the diagnosis of IBS, a food frequency consumption form for the last month will be used. This form consists of subgroups such as dairy products, meat-egg group, vegetables and fruits group, grain group, beverages, sugar/sweets/snacks group. Consumption frequency will be categorized as "never," "every day," "3-4 times a week," "1-2 times a week," "once in 15 days," and "once a month." Participants will also be questioned about whether the consumed foods cause gastrointestinal discomfort.

Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS) The Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS) will be used at the beginning and end of the study to assess the severity of symptoms of irritable bowel syndrome. To calculate symptom scores, participants will be asked 4 questions on a scale of 0 to 100. Based on the calculated score, the severity of the disease will be classified as follows: (0-74) for remission, (75-174) for mild, (175-299) for moderate, and (>300) for severe.

Quality of Life Scale in Irritable Bowel Syndrome Patients (IBS-QOL) The Irritable Bowel Syndrome Quality of Life Scale (IBS-QOL) will be applied at the beginning and end of the study to evaluate the level of quality of life of patients with irritable bowel syndrome. This questionnaire, designed for patients with irritable bowel syndrome, evaluates disease symptoms as well as the psychological, sociological effects of the disease, and its impact on individuals' sexual lives, among other topics. The questionnaire consists of 8 sub-scales, with 34 questions, allowing for the evaluation of quality of life on a scale of 100 points.

Visual Analog Scale (VAS-IBS) The Visual Analog Scale (VAS) is used to convert some non-numerically measurable values into numerical values. In this study, the VAS-IBS developed for patients with irritable bowel syndrome will be used. It consists of 10 questions and will be used at the beginning and end of the study. This scale includes evaluations such as abdominal pain, constipation, bloating/gas, nausea/vomiting, psychological state, and the impact of symptoms on daily life. Participants will mark their condition on a 100 mm line by indicating where their condition falls between the two extremes defined for each parameter (1: very poor, 10: very good). Additionally, participants will be asked to indicate whether they feel their bowels have completely emptied after using the toilet using this form.

Bristol Stool Form Scale To evaluate participants' stool forms at the beginning and end of the study, the Bristol Stool Form Scale will be used. This scale aims to estimate stool form based on 7 different stool shapes. It will be used at the beginning and end of the study. Improvement in stool form will be understood as approaching form number 4 on the scale.

Dietary Interventions Used for Medical Nutrition Therapy Two different types of diets will be used for a 4-week medical nutrition therapy intervention for participants in this study. These are a gluten-free diet and a low FODMAP diet. The low FODMAP diet involves the elimination of foods rich in fermentable oligo-, di-, monosaccharides and polyols, fructans, galactooligosaccharides (such as rye, barley, wheat, onions, and legumes), lactose-containing products (milk, yogurt, cheese), excessive fructose (apples, pears, watermelon, asparagus, honey), and foods rich in sorbitol, mannitol, and xylitol. It consists of a list indicating permitted and forbidden foods according to food groups. General recommendations are provided at the end of the diet list. The gluten-free diet is created by eliminating gluten-containing foods (such as wheat, barley, rye, etc.) from the diet. Permitted and forbidden foods are listed according to food groups, with general recommendations added at the end of the diet list. Participants will be provided with separate lists of permitted and forbidden foods for the low FODMAP diet and the gluten-free diet, along with general recommendations, and the diets will be explained to them. There will be no additional energy calculation or modified diet used in our study. Participants will be advised to prepare meals separately from household members and avoid forbidden foods for four weeks. Increasing the number of meals (5-6 meals) and avoiding gas-producing foods (cabbage, radish, legumes), carbon

ELIGIBILITY:
Inclusion Criteria:

* Participants between the ages of 18-65 who have been diagnosed with Irritable Bowel Syndrome (IBS) according to the Rome IV criteria,
* who are capable of making food choices independently,
* who do not have perception disorders or communication problems

Exclusion Criteria:

* Patients with inflammatory bowel disease
* celiac disease
* known lactose intolerance
* advanced cardiac, respiratory, renal, or hepatic diseases
* malignancy
* major psychiatric disorders, or a history of drug/alcohol abuse
* Patients with a history of previous abdominal surgery other than uncomplicated appendicitis
* pregnant and lactating patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-65 years
Enrollment: 75 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Food consumption records | To observe the effect of gluten free diet therapy on IBS quality of life after 1 month
  The gluten-free diet is created by eliminating gluten-containing foods (such as wheat, barley, rye, etc.) from the diet. Permitted and forbidden foods are listed according to food groups, with general recommendations added at the end of the diet list. Participants will be provided with separate lists of permitted and forbidden foods for the low FODMAP diet and the gluten-free diet, along with general recommendations, and the diets will be explained to them. There will be no additional energy calculation or modified diet used in our study.
Food consumption records | "To observe the effect of low FODMAP diet therapy on IBS quality of life after 1 month."
  The low FODMAP diet involves the elimination of foods rich in fermentable oligo-, di-, monosaccharides and polyols, fructans, galactooligosaccharides (such as rye, barley, wheat, onions, and legumes), lactose-containing products (milk, yogurt, cheese), excessive fructose (apples, pears, watermelon, asparagus, honey), and foods rich in sorbitol, mannitol, and xylitol. It consists of a list indicating permitted and forbidden foods according to food groups. General recommendations are provided at the end of the diet list.
Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS) | To observe the effect of diet therapy on GIS sypmtoms of life after 1 month."
  Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS) will be used at the beginning and end of the study to assess the severity of symptoms of irritable bowel syndrome. To calculate symptom scores, participants will be asked 4 questions on a scale of 0 to 100. Based on the calculated score, the severity of the disease will be classified as follows: (0-74) for remission, (75-174) for mild, (175-299) for moderate, and (>300) for severe.
Quality of Life Scale in Irritable Bowel Syndrome Patients (IBS-QOL) | To observe the effect of diet therapy on Quality of Life Scale of life after 1 month."
  The Irritable Bowel Syndrome Quality of Life Scale (IBS-QOL) will be applied at the beginning and end of the study to evaluate the level of quality of life of patients with irritable bowel syndrome. This questionnaire, designed for patients with irritable bowel syndrome, evaluates disease symptoms as well as the psychological, sociological effects of the disease, and its impact on individuals' sexual lives, among other topics. The questionnaire consists of 8 sub-scales, with 34 questions, allowing for the evaluation of quality of life on a scale of 100 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuh Naci Yazgan University, Kocasinan, Kayseri̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Research data will be shared as necessary.